CLINICAL TRIAL: NCT05163639
Title: Spinal Cord Associative Plasticity Study
Acronym: SCAP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Weill Medical College of Cornell University (Other); Bronx Veterans Medical Research Foundation, Inc (Other)
Responsible Party: Principal Investigator, Jason Carmel, Associate Professor, Columbia University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AAAT6563; 1R01NS124224-01 (NIH)
Record Dates: First submitted 2021-11-23; First posted 2021-12-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cervical Spinal Cord Injury; Tetraplegia/Tetraparesis; Cervical Myelopathy
Keywords: spinal cord injury; paired brain and spinal cord stimulation; convergent stimulation; spinal cord associative plasticity; transcutaneous spinal cord stimulation; intraoperative monitoring; upper-limb muscle activation; motor cortex; cervical spinal cord
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries | interventions — SREBP cleavage-activating protein

STUDY DESIGN:
Intervention Model Description: Participants with chronic SCI, participants with spondylotic radiculopathy or myelopathy scheduled to undergo elective cervical decompression surgery, and volunteers without neural injury will be prospectively enrolled in this interventional experimental study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 1. Uninjured participants - Immediate and lasting effects of non-invasive paired stimulation (Experimental): Participants will take part in the following to examine the immediate effects of combining cortical and spinal stimulation: A) Non-invasive pairing of cortical and spinal stimulation; B) Non-invasive repeated pairing of cortical and spinal stimulation (SCAP).
  Interventions: Procedure: Non-invasive pairing of cortical and spinal stimulation; Procedure: Non-invasive repeated pairing of cortical and spinal stimulation (SCAP)
- 2. Intraoperative participants - Immediate effects of paired stimulation (Experimental): Participants will take part in the following if they have been scheduled for a clinically indicated cervical surgery to examine the immediate effects of combining cortical and spinal stimulation: A) Non-invasive pairing of cortical and spinal stimulation; B) Intraoperative pairing of cortical and spinal stimulation.
  Interventions: Procedure: Non-invasive pairing of cortical and spinal stimulation; Procedure: Intraoperative pairing of cortical and spinal stimulation
- 3. Intraoperative participants - Lasting effects of SCAP (Experimental): Participants will take part in the following if they have been scheduled for a clinically indicated cervical surgery, to examine the lasting effects of repeated cortical and spinal stimulation: A) Non-invasive repeated pairing of cortical and spinal stimulation (SCAP); B) Intraoperative repeated pairing of cortical and spinal stimulation (SCAP).
  Interventions: Procedure: Non-invasive repeated pairing of cortical and spinal stimulation (SCAP); Procedure: Intraoperative repeated pairing of cortical and spinal stimulation (SCAP)
- 4. Chronic cervical SCI participants - Lasting effects of non-invasive SCAP (Experimental): Participants with chronic cervical SCI will take part in the following, to examine the lasting effects of repeated cortical and spinal stimulation: A) Non-invasive repeated pairing of cortical and spinal stimulation (SCAP).
  Interventions: Procedure: Non-invasive repeated pairing of cortical and spinal stimulation (SCAP)
- 5. Intraoperative participants - Lasting effects of SCAP at or below myelopathic region (Experimental): Participants will take part in the following if they have been scheduled for a clinically indicated cervical surgery, to examine the lasting effects of repeated cortical and spinal stimulation: A) Non-invasive repeated pairing of cortical and spinal stimulation (SCAP); B) Intraoperative repeated pairing of cortical and spinal stimulation (SCAP) at or below myelopathic region.
  Interventions: Procedure: Non-invasive repeated pairing of cortical and spinal stimulation (SCAP); Procedure: Intraoperative repeated pairing of cortical and spinal stimulation (SCAP) at or below myelopathic region

INTERVENTIONS:
Procedure: Non-invasive pairing of cortical and spinal stimulation — Transcranial magnetic stimulation (TMS) threshold, Transcutaneous spinal cord stimulation (TSCS) threshold, and peripheral and central motor conduction times will be determined. In the active intervention, two TMS pulse intensities will be tested: 90% and 120% of motor threshold. Two conditioning TSCS pulse intensities will be tested: 50% and 90% of response threshold. Single TSCS pulses will be delivered timed to arrive in the cervical spinal cord at a range of intervals from 30ms before to 30ms after the TMS pulse. The control conditions will include TMS only TSCS only and non-convergent pairing latency pairing stimulation.
  Arms: 1. Uninjured participants - Immediate and lasting effects of non-invasive paired stimulation; 2. Intraoperative participants - Immediate effects of paired stimulation
Procedure: Intraoperative pairing of cortical and spinal stimulation — The surgeon will position spinal cord electrodes on the epidural surface one level rostral (typically C4/C5) to the site of myelopathy. Spinal and cortical thresholds will be determined. Investigator will then test the immediate effects of paired stimulation by stimulating the cortex at 120% of threshold and the spinal cord at 90% of threshold at various latencies relative to the time of synchronous convergence. The control intervention will include cortical only (120%) spinal only (90%) and non-convergent latency pairing stimulation.
  Arms: 2. Intraoperative participants - Immediate effects of paired stimulation
Procedure: Non-invasive repeated pairing of cortical and spinal stimulation (SCAP) — Thresholds will be determined as above. Immediately prior to repetitive pairing, a set of 12 TMS pulses will be delivered at 120% threshold to measure the baseline cortical MEP. Likewise, a set of 12 TSCS pulses will be delivered at 120% of threshold to establish the baseline spinal MEP. For each session, baseline maximal pinch dynamometry will be determined. Immediately after the SCAP protocol is completed, response to TMS, TSCS, and maximal pinch dynamometry will be measured again every 10 minutes over the subsequent hour. The control conditions will include TMS only TSCS only and non-convergent pairing latency pairing stimulation.
  Arms: 1. Uninjured participants - Immediate and lasting effects of non-invasive paired stimulation; 3. Intraoperative participants - Lasting effects of SCAP; 4. Chronic cervical SCI participants - Lasting effects of non-invasive SCAP; 5. Intraoperative participants - Lasting effects of SCAP at or below myelopathic region
Procedure: Intraoperative repeated pairing of cortical and spinal stimulation (SCAP) — Intraoperative: Spinal and cortical thresholds will be determined. Immediately prior to repetitive pairing, a set of 12 baseline cortical pulses and 12 baseline spinal pulses will be delivered at 120% threshold. SCAP protocol will be applied, both of which have been successful at inducing lasting effects in the rat. After pairing, cortical stimulation at 120% of threshold and spinal cord stimulation at 120% threshold will be repeated every 10 minutes for the duration of surgery. In a subset of patients repeated pairing will be conducted with a latency that investigator does not expect will induce SCAP, or with electrodes placed over the ventral epidural surface. The control intervention will include repeated pairing at a non-convergent latency, as well as pairing of cortical stimulation with ventral epidural stimulation.
  Arms: 3. Intraoperative participants - Lasting effects of SCAP
Procedure: Intraoperative repeated pairing of cortical and spinal stimulation (SCAP) at or below myelopathic region — As per the intervention 'Intraoperative repeated pairing of cortical and spinal stimulation (SCAP)' targeted at or below myelopathic region.
  Arms: 5. Intraoperative participants - Lasting effects of SCAP at or below myelopathic region

SUMMARY:
Spinal cord associative plasticity (SCAP) is a combined cortical and spinal electrical stimulation technique developed to induce recovery of arm and hand function in spinal cord injury.

The proposed study will advance understanding of SCAP, which is critical to its effective translation to human therapy. The purpose of the study is to:

1. Determine whether signaling through the spinal cord to the muscles can be strengthened by electrical stimulation.
2. Improve our understanding of the spinal cord and how it produces movement.
3. Determine whether spinal surgery to relieve pressure on the spinal cord can improve its function.

Aim 1 is designed to advance mechanistic understanding of spinal cord associative plasticity (SCAP).

Aim 2 will determine whether SCAP increases spinal cord excitability after the period of repetitive pairing. In rats, SCAP augments muscle activation for hours after just 5 minutes of paired stimuli.

Whereas Aims 1 and 2 focused on the effects of paired stimulation in the context of uninjured spinal cord, Aim 3 assesses whether paired stimulation can be effective across injured cord segments. Aim 3 will incorporate the experiments from Aim 1 and 2 but in people with SCI, either traumatic or pre-operative patients with myelopathy in non-invasive experiments, or targeting myelopathic segments in intraoperative segments.

DETAILED DESCRIPTION:
For people with cervical spinal cord injury (SCI), regaining hand function is their highest priority. Currently there are no effective treatments for people living with paralysis or profound weakness after SCI. The goal of this project is to translate a promising therapy for improving arm and hand function after partial spinal cord injury to humans. The approach promotes repair of residual brain to spinal cord connections using combined motor cortex and spinal cord stimulation.

The direct brain to spinal cord connection is critical for skilled hand movement in health, and for the loss of movement after injury. After spinal cord injury, many nerve connections for movement are preserved. These connections can be strengthened by electrical stimulation.

The investigator has previously demonstrated that pairing brain and spinal cord stimulation strengthens spinal connections in rats. But it is unknown whether this is also applicable in humans. This study is designed to test this in people undergoing spine surgery for pain or decreased movement as well as non-invasively in people with traumatic spinal cord injury. There are three main goals of this project. First, the investigator will stimulate brain and spinal cord (intra-operatively and non-invasively) to try to study the influence of the timing of pairing brain and spinal cord stimulation. Second, the investigator will study how repeating the optimal timing (spinal cord associative plasticity; SCAP) will influence muscle responses over a longer period of time when relatively uninjured parts of the spinal cord are targeted. Finally, the investigator will study how the influence of this protocol changes when injured parts of the cord are targeted. Stimulation of brain and spinal cord intra-operatively will be performed with the same devices that maintain safety during the surgery, while non-invasive stimulation will be performed with non-significant risk devices.

Participants: Uninjured volunteers, individuals with chronic (> 1 year) cervical SCI, and individuals with cervical myelopathy or radiculopathy requiring clinically indicated decompressive surgery will be recruited. SCI and myelopathy participants will have partially retained motor function in the hand, scoring 1-4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction in left or right hand. Participants will also require detectable F-wave responses of the left or right abductor pollicis brevis (APB) to median nerve stimulation and/or first dorsal interosseous muscle (FDI) to ulnar nerve stimulation.

ELIGIBILITY:
NON-INVASIVE

Inclusion Criteria:

(All participants)

* Age between 18-80 years.
* Must have stable prescription medication for 30 days prior to screening
* Must be able to: abstain from alcohol, smoking and caffeine consumption on the day of each experiment; abstain from recreational drugs for the entirety of the study; commit to study requirements (i.e., 7 visits); provide informed consent.

(Able-bodied participants)

* No known central or peripheral neurological disease or injury.

(SCI participants - including patients scheduled for intraoperative procedures)

* Score of 1-4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction in left or right hand.

Exclusion criteria:

(All participants)

* Personal or extensive family history of seizures;
* Ventilator dependence or patent tracheostomy site;
* Use of medications that significantly lower seizure threshold, such as amphetamines, neuroleptics, dalfampridine, and bupropion;
* History of stroke, brain tumor, brain abscess, or multiple sclerosis;
* History of moderate or severe head trauma (loss of consciousness for greater than one hour or evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging);
* History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants in the head (except for inside mouth); cochlear implants; cardiac pacemaker/defibrillator; intracardiac lines; currently increased intracranial pressure; or other contraindications to brain or spine stimulation;
* Significant coronary artery or cardiac conduction disease; recent history of myocardial infarction and heart failure with an ejection fraction of less than 30% or with a New York Heart Association Functional Classification of Class III or IV;
* Recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg or diastolic pressure greater than 10 mm Hg, without rise in heart rate, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (this will be closely monitored during all screening and testing procedures);
* History of significant hearing problems;
* History of bipolar disorder;
* History of suicide attempt;
* Active psychosis;
* Recent history (>1 year) of chemical substance dependency or significant psychosocial disturbance;
* Heavy alcohol consumption (greater than equivalent of 5oz of liquor) within previous 48 hours;
* Open skin lesions over the face, neck, shoulders, or arms;
* Pregnancy; and
* Unsuitable for study participation as determined by study physician.

INTRA-OPERATIVE

Inclusion Criteria:

* Clinical indication for cervical spine surgery.

Exclusion criteria:

(For experiments involving cortical stimulation)

* Epilepsy;
* A history of skull surgery with metal implants;
* Cochlear implants;
* Patients with aneurysm stents in neck or brain blood vessels;
* Evidence of skull shrapnel; (For experiments involving spinal cord stimulation)
* Stimulation devices in the neck or chest (e.g., vagal nerve stimulation, cardiac patients with pacemakers)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Size of hand muscle response to brain stimulation during combined brain and spinal stimulation | Immediate
  Size of hand muscle response will be measured in response to brain and spinal cord stimulation timed to converge in the spinal cord. This value will be normalized to the muscle response for brain only stimulation. This applies to Arms 1-2.
Size of hand muscle response to brain stimulation after SCAP | Immediately after SCAP
  Size of hand muscle response will be measured in response to brain and spinal cord stimulation timed to converge in the spinal cord. This value will be normalized to the equivalent measure taken before the SCAP protocol. This applies to Arms 3-5.

SECONDARY OUTCOMES:
Size of hand muscle response to spinal cord stimulation | Immediately after SCAP
  Size of hand muscle response will be measured in response to brain and spinal cord stimulation timed to converge in the spinal cord. This value will be normalized to the equivalent measure taken before the SCAP protocol.
Duration of effect of SCAP on subsequent responses to brain or spinal cord stimulation | 1 hour after SCAP
  Time taken for the size of hand muscle response to fall to 50% of its maximal post-SCAP level.
Pinch force | Immediately after SCAP
  Pinch opposition strength between the tips of the thumb and third finger (a task highly dependent on cortical transmission to C8-T1 spinal circuitry will be measured using a handheld dynamometer. Force and root mean square (RMS) of electromyographic activity will be recorded. Maximal pinch dynamometry will be compared to baseline measurement.
Amplitudes of H-reflex ratio | Immediately after SCAP
  H-reflex amplitudes (Hmax/Mmax), a biomarker for spasticity triggered with 1.0 ms pulses over the median nerve at the elbow.
Threshold for triggering muscle response from brain stimulation | Immediately after SCAP
  The threshold for transcutaneous cortical electrical stimulation will be measured by increasing the voltage from 50V in 50V steps, until a MEP is detected.
Threshold for triggering muscle response from spinal cord stimulation | Immediately after SCAP
  The threshold for spinal cord stimulation will be measured by increasing the stimulation amplitude from 1mA in 1mA steps, until an evoked potential is observable in the target muscle, or our safety limit is reached. In cases where clear evoked responses cannot be generated within stimulation amplitude safety limits, 3 pulse stimuli will be used, or investigator will modify target muscle for the remainder of the experiment. Study will target APB, but more responsive muscles may be substituted.
Size of hand muscle response to spinal cord stimulation (lasting) | 30 minutes after SCAP
  Size of hand muscle response will be measured in response to brain and spinal cord stimulation timed to converge in the spinal cord. This value will be normalized to the equivalent measure taken before the SCAP protocol.
Pinch force (lasting) | 30 minutes after SCAP
  Pinch opposition strength between the tips of the thumb and third finger (a task highly dependent on cortical transmission to C8-T1 spinal circuitry will be measured using a handheld dynamometer. Force and root mean square (RMS) of electromyographic activity will be recorded. Maximal pinch dynamometry will be compared to baseline measurement.
Amplitudes of H-reflex ratio (lasting) | 30 minutes after SCAP
  H-reflex amplitudes (Hmax/Mmax), a biomarker for spasticity triggered with 1.0 ms pulses over the median nerve at the elbow.
Threshold for triggering muscle response from brain stimulation (lasting) | 30 minutes after SCAP
  The threshold for spinal cord stimulation will be measured by increasing the stimulation amplitude from 1mA in 1mA steps, until an evoked potential is observable in the target muscle, or our safety limit is reached. In cases where clear evoked responses cannot be generated within stimulation amplitude safety limits, 3 pulse stimuli will be used, or investigator will modify target muscle for the remainder of the experiment. Study will target APB, but more responsive muscles may be substituted.

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Carmel, M.D., Ph.D., Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Bronx Veterans Medical Research Foundation, Inc, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, individual-level data will be deposited to appropriate public repositories, such as Open Data Commons for Spinal Cord Injury (https://scicrunch.org/odc-sci), Figshare, or others.
  This will allow more powerful meta-analysis of disparate smaller studies, a need which is even more urgent in neurorehabilitation than in other fields that are more amenable to large drug studies.
Supporting Information: Study Protocol, SAP
Time Frame: Within 6 months of manuscript preparation.
Access Criteria: Individually identifiable data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions described in the authorization and consent.
  A Data Use Agreement (DUA) will indicate adherence to any applicable Informed Consent provisions, and prohibits the recipient from identifying or re-identifying any individual whose data are included in the dataset.